CLINICAL TRIAL: NCT05977842
Title: Drug-coated Balloon in de Novo Chronic Total Occlusions (CTO-DENOVO Registry)
Brief Title: Drug-coated Balloon in de Novo Chronic Total Occlusions
Acronym: CTO-DENOVO
Status: Completed | Type: Observational
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: CTO-DENOVO
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-10

CONDITIONS: Coronary Artery Disease; Total Occlusion of Coronary Artery
Keywords: chronic total occlusion; percutaneous coronary intervention; drug-coated balloon
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CTO PCI using DCB-only strategy — Successful CTO recanalization treated with DCB at the occlusion site

SUMMARY:
The CTO-DENOVO study is a multicenter registry of consecutive patients with de novo coronary chronic total occlusions (CTO) undergoing successful CTO recanalization with the use of drug-coated balloon (DCB)-only strategy. The primary endpoint is target lesion failure at 6 months. The secondary endpoints are: 1) late lumen loss on follow-up angiography, and 2) minimal lumen area on follow-up intravascular ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* de novo coronary CTO undergoing successful recanalization with the use of DCB-only strategy at the occlusion site

Exclusion Criteria:

* de novo coronary CTO undergoing successful recanalization with the use of DES at the occlusion site
* in-stent CTO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with de novo CTO undergoing successful PCI with the use of DCB-only strategy.
Sampling Method: Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2012-12-15 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | 6 months
  Composite of cardiac death, target vessel-related myocardial infarction, or clinically-driven target lesion revascularization

SECONDARY OUTCOMES:
Late lumen loss | 3 months
  In-segment late lumen loss on follow-up angiography (in-segment equals DCB plus the proximal and distal 5-mm margins)
Minimal lumen area | 3 months
  In-segment minimal lumen area on follow-up intravascular ultrasound (IVUS) (in-segment equals DCB plus the proximal and distal 5-mm margins)

CONTACTS AND LOCATIONS:
Overall Officials: Maksymilian Opolski, MD, Principal Investigator — National Institute of Cardiology
Locations (35):
- Austria (2):
  - Graz University Heart Center, Graz
  - Klinik Ottakring, Vienna
- Jolimont Hospital, Uccle, Belgium
- Županijska bolnica Čakovec, Čakovec, Croatia
- Czechia (3):
  - University Hospital Brno, Brno
  - Liberec Regional Hospital, Liberec
  - Kardiologické Centrum AGEL, Pardubice
- Lille University Hospital, Lille, France
- Hospital zum Heiligen Geist, Kempen, Germany
- Hungary (2):
  - University of Debrecen, Debrecen
  - University of Szeged, Szeged
- Shamir Assaf Harofeh MC, Be’er Ya‘aqov, Israel
- Italy (3):
  - Humanitas University, Milan
  - Villa Sofia Hospital, Palermo
  - Santissima Annunziata Hospital, Savigliano
- Poland (17):
  - Medical University of Bialystok, Bialystok
  - American Heart of Poland, Bielsko-Biala
  - John Paul II Western Hospital, Grodzisk Mazowiecki
  - Jagiellonian University Medical College, Krakow
  - John Paul II Hospital, Krakow
  - MSWiA Hospital, Lodz
  - 1st Military Hospital, Lublin
  - MSWiA Hospital, Lublin
  - Poznan University of Medical Sciences, Poznan
  - SP ZOZ Hospital, Puławy
  - MSWiA Hospital, Rzeszów
  - Bielanski Hospital, Warsaw
  - Military Institute of Medicine, Warsaw
  - National Institute of Cardiology, Warsaw
  - Dr Alfred Sokolowski Specialist Hospital, Wałbrzych
  - Wroclaw Medical University, Wroclaw
  - Silesian Center for Heart Disease, Zabrze
- Romania (2):
  - Heart Institute, Cluj-Napoca
  - Emergency Clinical County Hospital, Oradea
- Hospital Clínico Universitario de Valladolid, Valladolid, Spain